CLINICAL TRIAL: NCT01202929
Title: Correlation of High Resolution Esophageal Manometry With Symptoms
Status: Withdrawn | Type: Observational
Why Stopped: Principal investigator has left the Institution
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Other Study IDs: 10.0057
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Achalasia; Dysphagia; GERD; Chest Pain; Post Fundoplication
Keywords: High Resolution Manometry; achalasia; dysphagia; GERD; chest pain; Post fundoplication
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders; Gastroesophageal Reflux; Chest Pain | interventions — Manometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Type I achalasia: classic achalasia: complete esophageal motor failure
  Interventions: Procedure: High Resolution Manometry
- Type II achalasia: compression achalasia: simultaneous panesophageal pressurization with aperistalsis
  Interventions: Procedure: High Resolution Manometry
- Type III achalasia: spastic achalasia with aperistalsis: 100% spasm
  Interventions: Procedure: High Resolution Manometry

INTERVENTIONS:
Procedure: High Resolution Manometry — High Resolution Manometry which uses 36 solid state sensors spaced at 1-cm intervals, positioned from the hypopharynx to the stomach.
  Other Names: Manometry; Achalasia

SUMMARY:
High Resolution Manometry is a new technology that utilizes 36 solid state sensors on a thin catheter spaced at 1-cm intervals. One can more effectively measure the pressure of the esophagus. It includes a sophisticated software to display the pressures data as color topography plot using time, length of the esophagus and pressure within the entire esophagus. It is unclear if this technology improvement actually correlates with patient's symptoms.

DETAILED DESCRIPTION:
In a 2007 retrospective study performed using this technology, 400 subjects referred to the motility lab underwent high resolution manometry (HRM) for complaints of dysphasia, gastroesophageal reflux disease, chest pain and miscellaneous complaints. HRM offered greater detail of individual contracting segments of the esophagus, including the duration of contraction and propagation of individual contractions.

For example, a new subclass of achalasia was defined by HRM. In this classification, achalasia is divided into types 1, 2 and 3. Type 1 corresponds to classic achalasia (complete esophageal motor failure), type 2 is a compression achalasia (simultaneous panesophageal pressurization with aperistalsis), and type 3 is spastic achalasia with aperistalsis (100% spasm). However, it is unclear if this categorization represents a spectrum of disease among patients with achalasia, or it represents distinct subgroups of patients with different symptom presentation and etiology.

This study will attempt to correlate the data from HRM to patient's chief compliants, symptom severity, and clinical presentation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are referred to the motility lab to undergoing esophageal HRM for various clinical indications.

Exclusion Criteria:

* Pregnancy
* Unable to give consent
* Less than 18 years old
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from patients referred to the University Medical Associates motility lab for high resolution manometry
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Differences and similarities in patients with achalasia | at 24 months
  To determine the differences and similarities in the clinical presentation of patients with type 1, 2 and 3 achalasia based on the Chicago classification for HRM

SECONDARY OUTCOMES:
Esophageal dysmotility in patients with dysphagia and GERD symptoms | at 24 months
  To determine the prevalence of esophageal dysmotility using the Chicago classification based on primary chief complaints.
HRM parameters | at 24 months
  To determine if HRM parameters reflect esophageal physiology between contractile strength of the esophagus and GEJ residual pressure obstructing esophageal flow.
Esophageal dysmotility in patients with postfundoplication compliants | at 24 months
  To determine the prevalence of esophageal dysmotility using the Chicago classification based in patients with postfundoplication complaints.
Correlation between HRM and symptoms | At 24 months
  To determine if HRM parameters reflect symptom presentations.

CONTACTS AND LOCATIONS:
Overall Officials: John Wo, MD, Principal Investigator — University of Louisville School of Medicine
Locations (1):
- University of Louisville, Louisville, Kentucky, United States